CLINICAL TRIAL: NCT04339946
Title: Bidimensional Rectal-water Contrast-transvaginal Ultrasonography (2D-RWC-TVS) Versus 3D-RWC-TVS in the Diagnosis of Rectosigmoid Endometriosis
Acronym: 3Dvs2D-RWC-TVS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal investigator, Ospedale Policlinico San Martino
Other Study IDs: 3Dvs2D-RWC-TVS
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis, Rectum; Endometriosis of Colon
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspicious of rectosigmoid endometriosis
  Interventions: Diagnostic Test: Three-dimensional rectal water contrast transvaginal ultrasonography (3D-RWC-TVS); Diagnostic Test: Two-dimensional rectal water contrast transvaginal ultrasonography (2D-RWC-TVS)

INTERVENTIONS:
Diagnostic Test: Three-dimensional rectal water contrast transvaginal ultrasonography (3D-RWC-TVS) — Rectal water contrast transvaginal ultrasonography is based on the distention of rectosigmoid with saline solution. Three-dimensional reconstructions convert standard 2D grayscale ultrasound acquisitions into a volumetric dataset.
Diagnostic Test: Two-dimensional rectal water contrast transvaginal ultrasonography (2D-RWC-TVS) — Rectal water contrast transvaginal ultrasonography is based on the distention of rectosigmoid with saline solution.

SUMMARY:
An accurate diagnosis of the presence, location and extent of the rectosigmoid endometriosis is of paramount importance for the clinicians in order to inform the patients on the potential surgical or medical treatments. It is well established that transvaginal ultrasonography is the first-line investigation in patients with suspicion of deep infiltrating endometriosis.

An improvement in the performance of transvaginal ultrasonography in diagnosing rectosigmoid endometriosis may be obtained by using rectal water contrast during transvaginal ultrasonographic scan.

ELIGIBILITY:
Inclusion Criteria:

* pain and intestinal symptoms suggestive of rectosigmoid endometriosis

Exclusion Criteria:

* previous surgical diagnosis of intestinal endometriosis
* previous radiological diagnosis of intestinal endometriosis (based on Magnetic Resonance or double-contrast barium enema)
* history of colorectal surgery (except appendectomy)
* contraindications to bowel preparation or computed colonography (such as non-compliant patients and rectal malformations)
* previous bilateral ovariectomy
* psychiatric disorders

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with clinical presentation suspected for rectosigmoid endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
To compare the accuracy of 3D-RWC-TVS and 2D-RWC-TVS in the diagnosis of rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

SECONDARY OUTCOMES:
To compare the precision of 3D-RWC-TVS and 2D-RWC-TVS in estimating the length (mid-sagittal diameter) of the rectosigmoid endometriotic nodules | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the accuracy of 3D-RWC-TVS and 2D-RWC-TVS in the diagnosis of multifocal rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the precision of 3D-RWC-TVS and 2D-RWC-TVS in estimating and the distance between the lower margin of the rectosigmoid endometriotic nodules and the anal verge | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the precision of 3D-RWC-TVS and 2D-RWC-TVS in estimating rectosigmoid lumen stenosis due to endometriotic nodule | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morotti M, Ferrero S, Bogliolo S, Venturini PL, Remorgida V, Valenzano Menada M. Transvaginal ultrasonography with water-contrast in the rectum in the diagnosis of bowel endometriosis. Minerva Ginecol. 2010 Jun;62(3):179-85. English, Italian. PMID 20595942